CLINICAL TRIAL: NCT03751501
Title: Photocoagulation of Capillary Macro-aneurysms in Addition to the Standard Treatment of Macular Edema Due to Diabetic Retinopathy. "TaLa_DME"
Brief Title: Targeted Laser in Diabetic Macular Edema
Acronym: TaLa-DME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P18-01
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-12

CONDITIONS: Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized into one of the 2 study arms groups: "standard of care" group with sham laser or experimental group with laser.
  Both group with laser or sham laser will be performed in combination with anti VEGF treatment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Indocyanine green-Guided Targeted Laser photocoagulation combines routine procedures, that are, the detection of macro-aneurysms by ICG angiography, laser photocoagulation and optional post-laser verification of the effectiveness of the photothrombosis by OCT. Indocyanine green-Guided Targeted Laser photocoagulation is administered in combination with anti VEGF treatment
  Interventions: Procedure: Indocyanine green-Guided Targeted Laser photocoagulation
- Control Group (Sham Comparator): Sham laser is administered at randomization visit and repeated if needed 3 month later in combination with anti VEGF treatment
  Interventions: Procedure: Sham laser

INTERVENTIONS:
Procedure: Indocyanine green-Guided Targeted Laser photocoagulation — Detection of macro-aneurysms by ICG angiography, laser photocoagulation and optional post-laser verification of the effectiveness of the photothrombosis by OCT.
  Arms: Experimental Group
Procedure: Sham laser — Therapeutic procedure used in ophthalmology
  Arms: Control Group

SUMMARY:
Our hypothesis is that implementing laser photocoagulation (IGTL) as an adjunctive treatment to intravitreal injections should lead to a significant reduction in the need for intravitreal injections in patients with diabetic macular edema without adverse consequences for visual acuity.

DETAILED DESCRIPTION:
This study will be French, multicenter parallel group, 2-arms, randomized, sham laser-controlled, double-blind trial evaluating the effect of IGTL as an adjunctive procedure to intravitreal injections in patients with DME.

Acts which are the subject of the study: indocyanine green-Guided Targeted Laser photocoagulation (IGTL): this combines routine procedures, that are, the detection of macro-aneurysms by ICG angiography, laser photocoagulation and optional post-laser verification of the effectiveness of the photothrombosis by OCT.

Study act: the treatment study includes a baseline laser treatment (experimental group) or sham laser (control group) at randomization, repeated if needed 3 month later, administered in combination with anti VEGF treatment, consisting of 3 monthly injections in the first 3 months, and a maintenance phase with monthly visits where retreatment is administered as needed through a PRN regimen, based on morphological (retinal thickness on OCT) and functional (visual acuity) criteria.

To evaluate the interest of IGTL in real conditions, the choice of the anti VEGF treatment used for intravitreal injection (Ranibizumab or Aflibercept, which have French marketing authorizations) is left to each investigator (equivalent therapeutic efficacy). Bevacizumab is ruled out due to its lower efficacy compared with Aflibercept among eyes with worse baseline VA, that represent the majority of the patients in our study. In addition, bevacizumab is currently off-label in France for DME If both eyes are eligible at the time of randomization, only one eye will be included and analyzed. However, the fellow eye will be treated with the randomization-assigned treatment and the testing will be performed on each eye.

Risks and constraints involved in the study: these procedures are commonly done in ophthalmology care settings; no additional risk is expected due to the study.

Expected benefits for the participants and for the company: These procedures are commonly done in ophthalmology care settings; no additional risk is expected due to the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic women and men ≥18 years
* with visual acuity lower or equal than 20/32 ( ≤ 74 TaLaDME protocol_v1.2_12.07.2018 9/76 ETDRS letters)
* with central retinal thickness of more than 300μm in Spectral Domain OCT (SD-OCT) and/or presence of retro-foveal hard exudates
* due to DME
* with one or more macro-aneurysms with a diameter greater than 150 μm in the posterior pole
* with health insurance
* who signed the written informed consent form

Exclusion Criteria:

* Presence of age-related drusens or of a macular degeneration in one or both any eyes
* Significant opacity of the ocular media that could contribute to decreased visual acuity
* macro-aneurysm(s) mainly responsible for the DME located less than 500μm from the center of the fovea (i.e. within 1 disc radius of the fovea),
* Steroids injection within the last 4 months
* proliferative diabetic retinopathy requiring panretinal photocoagulation or associated with posterior tractional retinal detachment that may be worsened by the use of anti-VEGF therapy
* myocardial infarction or stroke within the last 3 months
* Cataract surgery within the last 3 months
* Local treatment with prostaglandin
* Women who are pregnant, breast feeding or of child bearing age without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Number of anti VEGF injections | 12months
  as measured between baseline and M12
Change in Visual Acuity (Letters) | 12 months
  As measured by the Early Treatment Diabetic Retinopathy Study (ETDRS)

SECONDARY OUTCOMES:
Change in central macular thickness | 12 months
  as measured between baseline and M12
Cost of treatment | 12 months
  as measured between baseline and M12
Incremental cost-utility ratio | 12 months
  as measured between baseline and M12
Impact on quality of life using standard score evolution | 12 months
  as measured between baseline and M12
Number of AEs/SAEs | 36 months
  as measured between baseline and M36

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, PU-PH, Principal Investigator — Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France

REFERENCES:
- [Derived] Dupas B, Castro-Farias D, Girmens JF, Eginay A, Couturier A, Villeroy F, Delyfer MN, Creuzot-Garcher C, Giocanti-Auregan A, Beral L, Arndt C, Mesnard C, Vicaut E, Chaumet-Riffaud P, Durand-Zaleski I, Paques M. Photocoagulation or sham laser in addition to conventional anti-VEGF therapy in macular edema associated with TelCaps due to diabetic macular edema or retinal vein occlusion (TalaDME): a study protocol for a multicentric, French, two-group, non-commercial, active-control, observer-masked, non-inferiority, randomized controlled clinical trial. Trials. 2024 Apr 22;25(1):273. doi: 10.1186/s13063-024-07994-1. PMID 38649937